CLINICAL TRIAL: NCT06532214
Title: Clinical Retrospective Study Analysis of Postoperative Complications Following Hepatectomy
Status: Recruiting | Type: Observational
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: NFEC-2023-245
Record Dates: First submitted 2024-07-29; First posted 2024-08-01 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Liver Failure; Liver Dysfunction
Keywords: hepatectomy; liver failure; Post-hepatectomy liver failure
MeSH Terms: conditions — Liver Failure; Liver Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- PHLF/NPHLF: PHLF:Post-hepatectomy liver failure,PHLF is commonly diagnosed and classified according to the criteria of the International Study Group for Liver Surgery (ISGLS), utilizing markers of liver function measured on or after postoperative day 5 (POD5). NPHLF:Patients who did not experience liver failure following hepatectomy.
  Interventions: Diagnostic Test: International Study Group for Liver Surgery (ISGLS)
- Liver Cirrhosis/No Liver Cirrhosis: Whether the patient has cirrhosis

INTERVENTIONS:
Diagnostic Test: International Study Group for Liver Surgery (ISGLS) — According to the ISGLS criteria, the patient was judged to have liver failure and further analysis
  Groups: PHLF/NPHLF

SUMMARY:
Hepatectomy is a crucial surgical method for treating liver diseases such as liver cancer, hepatic hemangiomas, and biliary stones. Although hepatectomy has achieved significant therapeutic effects, postoperative complications remain an inevitable issue. Complications following hepatectomy include liver failure, hepatic vascular thrombosis, wound infection at the hepatic incision, and bile leakage, among others. These complications pose a serious threat to patients' health and life, and also increase the waste of medical resources and the cost of treatment. Currently, research on postoperative complications of hepatectomy mainly focuses on small sample studies from a single center, and most studies only focus on a specific complication, lacking comprehensive and systematic analysis. Therefore, it is necessary to conduct a retrospective study analysis of complications related to hepatectomy to more comprehensively and objectively understand the incidence, risk factors, prevention, and treatment of postoperative complications, providing clinical doctors with more scientific treatment plans and guidance.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients aged 18-80 years 2.Patients who underwent liver resection surgery at the participating centers

Exclusion Criteria:

* Exclusion criteria are as follows:

  1. Prior cancer treatments such as transarterial chemoembolization, ablation, or targeted therapy.
  2. Repeat liver resection surgeries.
  3. Presence of other malignancies.
  4. Concurrent end-stage diseases including active infections, respiratory failure, decompensated heart failure, and autoimmune disease exacerbations.
  5. Inadequate clinical data availability in medical records.

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients who underwent liver resection surgery at the participating centers
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Post-hepatectomy liver failure (PHLF) | On and after the 5th postoperative day
  PHLF is commonly diagnosed and classified according to the criteria of the International Study Group for Liver Surgery (ISGLS), utilizing markers of liver function measured on or after postoperative day 5 (POD5).

SECONDARY OUTCOMES:
mortality | During 30 days after surgery
  The patient died postoperatively

CONTACTS AND LOCATIONS:
Locations (1):
- Nanfang Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided
To ensure the protection of patients' clinical information data, ethical committee approval is required before sharing data with other research studies. This process is crucial for maintaining patient confidentiality and adhering to privacy regulations and ethical standards in research.

REFERENCES:
- [Derived] Wang K, Yang Q, Li K, Tang S, Zhang B, Liao X, Du S, Fu W, Li Z, Chen H, Xie H, Huang P, Li J, Wang Q, Liu H, Huang Z, Heng PA, Wan X, Li C, Si W. Learning-based early detection of post-hepatectomy liver failure using temporal perioperative data: a nationwide multicenter retrospective study in China. EClinicalMedicine. 2025 May 6;83:103220. doi: 10.1016/j.eclinm.2025.103220. eCollection 2025 May. PMID 40630620